CLINICAL TRIAL: NCT02785497
Title: Electrical Stimulation of Cutaneous Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, PHD Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1143-6541
Record Dates: First submitted 2013-05-28; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Ulcer; Burns
Keywords: Electrical stimulation; wound healing; Polarity current; Burn; Chronic ulcer
MeSH Terms: conditions — Burns | interventions — Control Groups; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Chronic ulcer patients will be treated with 50 minutes of the high-voltage current or 10 minutes of the diadynamic current. To burn patients 50 minutes high voltage current in the donor area. For both group the metal electrodes will be sterilized and the negative polarity in the active electrode.
  50 min, 100Hz, intensity according to the sensitivity patient - High Voltage; 10 min, intensity according to the sensitivity patient - Diadynamic
  Interventions: Other: Treatment group
- Control group (Sham Comparator): For the control group the unit is turned on, the time will pass but will not be given intensity
  50min, 100Hz, Intensity according to the sensitivity patient
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — will be turn on the equipment, positioning the patient but no put intensity
  Other Names: Sham group
  Arms: Control group
Other: Treatment group — This group will receive electrostimulation
  Other Names: Electrical stimulation; polar current; Current treatment; current stimulation
  Arms: Treatment group

SUMMARY:
Skin lesions, such as chronic ulcers and burns, represent a serious public health problem due to high government costs, and scarce successful conservative treatments.There is a growing scientific literature on the use of electrotherapy in the process of wound healing, but in return there is a dearth of scientific studies on the use of various types of currents and the different parameters in the proposed treatments.

DETAILED DESCRIPTION:
This project proposes the use of polarized currents to increase the speed of healing in chronic ulcers and donor sites in burn patients. Will be included 30 patients with chronic ulcers and 30 burn patients undergoing skin graft surgery, will be randomized into control and treated groups. For the ulcer chronic group treatment will be with 50 minutes high voltage and 10 minutes diadynamica current and the burn group only 50 minutes high voltage current.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the rehabilitation center of Clinical Hospital with chronic ulcer, Faculty of Medicine of Ribeirão Preto / USP, in the period between january 2010 and december 2011
* all patients admitted to the Burns Unit of Clinical Hospital, Faculty of Medicine of Ribeirão Preto / USP, in the period between march 2011 and december 2012

Exclusion Criteria:

* Infection
* weight below 16kg

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
clinical evaluation of the lesion | Two years
  will be documented appearance of the wound

SECONDARY OUTCOMES:
standard photographic records of the wounds and quantification by digital software | Two years
  Assessment the wound area image for image j software and validate CAPAS software for the healing wound image by descriptors textures

OTHER OUTCOMES:
Expert in evaluating healing images for a score | Two years
  Assessment to validate score in injury healing cutaneous

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Guirro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br